CLINICAL TRIAL: NCT01996189
Title: Arterial Puncture Using Insulin Syringe is Less Painful Than Standard Syringe, a Randomized Crossover Study
Brief Title: Arterial Puncture Using Insulin Syringe is Less Painful Than Standard Syringe
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Emergency, Doctor, National University Hospital, Singapore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: JPFF-11-1-YYW
Record Dates: First submitted 2013-10-28; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Insulin Infusion Systems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin (Experimental): Arterial puncture with an insulin syringe followed by arterial puncture with standard needle.
  Interventions: Device: Standard needle BBraun Sterican® 23G and 25mm in length; Device: Insulin
- Standard (Active Comparator): Arterial puncture with standard needle followed by arterial puncture with insulin syringe.
  Interventions: Device: Standard needle BBraun Sterican® 23G and 25mm in length; Device: Insulin

INTERVENTIONS:
Device: Standard needle BBraun Sterican® 23G and 25mm in length — Arterial puncture using the hypodermic needle (BBraun Sterican® 23G and 25mm in length) attached to a 3 ml syringe.
Device: Insulin — Arterial puncture using the insulin syringe (Terumo®- 0.5 ml with attached needle 29G and 13mm in length)

SUMMARY:
The primary objective is to compare the difference in the pain score in radial arterial puncture using the insulin needle versus the standard 23G hypodermic needle.

DETAILED DESCRIPTION:
In a randomised, crossover design, healthy volunteers were recruited to receive bilateral radial arterial punctures. They were assigned to receive either the insulin or the standard needle as the first puncture using block randomisation. The primary outcome was the pain score measured on a 100mm visual analogue scale (VAS) and the secondary outcomes were procedural complications and rate of haemolysis.

ELIGIBILITY:
Inclusion Criteria:

* age above 21

Exclusion Criteria:

* concurrent antipyretic use in the last 24 hrs,
* presence of painful conditions eg fracture, rheumatoid arthritis
* history of peripheral vascular disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) score in millimetres | Immediately after each puncture ( average within 5 minutes)
  Immediately following the radial arterial punctures the outcome assessor asked the volunteer to assess the discomfort that was caused by the puncture. The volunteer was asked to place a slash on a 100 mm VAS sheet. The VAS showed "no pain" at 0 mm and "worst pain" at 100 mm.

SECONDARY OUTCOMES:
blood haemolysis | Immediately after collection
  The serum collected during the punctures was analysed for the amount of free haemoglobin. We define presence of haemolysis as free haemoglobin concentration of more than 100 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Irwani Ibrahim, MBBS, Principal Investigator — National Unversity Health Systems; Yau Ying Wei, MBBS, Principal Investigator — National University Health Systems
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore